CLINICAL TRIAL: NCT06551688
Title: Influence of Preoperative Vitamin D Level on Postoperative Pain in Breast Cancer Surgery Patients: A Prospective Observational Study
Brief Title: Influence of Preoperative Vitamin D Level on Postoperative Pain in Breast Cancer Surgery Patients
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Hamed, Associate professor of anaesthesiology, Fayoum University
Other Study IDs: D328
Record Dates: First submitted 2024-07-03; First posted 2024-08-13 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Cancer Breast; Hypovitaminosis D
Keywords: preoperative vitamin D level; postoperative pain; cancer breast surgery
MeSH Terms: conditions — Breast Neoplasms; Vitamin D Deficiency; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group D: vitamin D-deficient group (<30nmol/L)
  Interventions: Diagnostic Test: Serum 25(OH)D level
- group S: vitamin D-sufficient group (≥30nmol/L)
  Interventions: Diagnostic Test: Serum 25(OH)D level

INTERVENTIONS:
Diagnostic Test: Serum 25(OH)D level — The characteristics of 25 (OH) D3 are relatively longer half-life than 1.25 (OH)2 D3, stability, strong detection repeatability, and no biological activity. Generally, systemic levels of the more stable 25 (OH) D3 are considered to be the best index to reflect status of vitamin D in the individual patient

SUMMARY:
Vitamin D deficiency is a general problem that vigorously affects human health . Breast cancer is the most frequently diagnosed life-threatening cancer in women and the leading cause of cancer death among women.Vitamin D deficiency is common in breast cancer patients and some evidence suggests that low vitamin D status enhances the risk for disease development or progression .

Though the relationship between vitamin D and breast cancer is unclear . Several research studies currently support vitamin D deficiency as a risk factor for breast cancer. Observational studies have also revealed significant relationships of vitamin D with breast cancer, colorectal cancer, prostate cancer and pancreatic cancer .

However, no work has been done to investigate the relationship between vitamin D deficiency and acute postoperative pain in breast cancer surgery patients. In the current study we will investigate the relationship between preoperative vitamin D levels and acute postoperative pain in cancer breast surgery patients.

The aim of current study is to investigate the relationship between preoperative vitamin D levels and acute postoperative pain in breast cancer surgery patients.

DETAILED DESCRIPTION:
This study will be performed in the FAYOUM University Hospital after the local Institutional Ethics Committee and local institutional review board approval. Newly diagnosed and pathologically proven breast cancer patients who are prepared for elective breast cancer surgery will be recruited from the general surgery department of our hospital. The study design will be prospective observational study. A detailed informed consent will be signed by the eligible patients before recruitment.

Measurement of vitamin D:

The characteristics of 25 (OH) D3 are relatively longer half-life than 1.25 (OH)2 D3, stability, strong detection repeatability, and no biological activity. Generally, systemic levels of the more stable 25 (OH) D3 are considered to be the best index to reflect status of vitamin D in the individual patient .

study design:

Serum 25(OH)D levels will be measured preoperative . Patients will be divided into two groups :

(1) group D: vitamin D-deficient group (<30nmol/L); and (2) group S: vitamin D-sufficient group (≥30nmol/L) .

Randomization:

Preoperative serum 25(OH) D levels will be assessed by an anaesthesiologist who will not be included in the study, to get the number of patients required in each group. Randomization will be done via computer-generated random numbers that will be placed in separate closed envelopes and will be opened by study investigators just after induction of general anaesthesia. Neither the patients, the study investigators, the attending clinicians nor the data collectors will be aware of the allocation of groups till the study ends. The patients will be allocated in 1:1 ratio to one of the two groups: group D: vitamin D-deficient group (n= 92 ), and group S: vitamin D-sufficient group (n= 92).

Anaesthesia procedure:

All patients will undergo routine preoperative investigations; CBC, coagulation profile, liver function tests, kidney function tests, ECG and preoperative serum 25(OH)D level. Upon arrival to the operating room, standard monitors (5-lead electrocardiogram, pulse oximeter, noninvasive blood pressure monitoring) will be applied and continue all over the operation. An IV access will be established. All patients will receive IV ondansetron 4 mg before induction of anesthesia as a premedication. General anesthesia will be performed as follows: induction using IV propofol (2mg/kg), atracurium (0.5mg/kg), and fentanyl (1 microgram/kg). A cuffed endotracheal tube (7mm ID) will be placed to secure the airway. Mechanical ventilation parameters will be adjusted to ensure proper oxygenation and ventilation with normocapnia. Maintenance of anesthesia will be made using inhalational anesthesia with isoflurane 1.5% volume concentration and IV atracurium (0.1 mg/kg) every 20 minutes. Continuous hemodynamic monitoring of blood pressure and heart rate will be done . If the systolic blood pressure decreased to a 20% below the baseline or less than 90 mmHg, 5 mg of ephedrine will be injected IV. Moreover, if the heart rate reduced to a 50 bpm or less, 0.5 mg of atropine will be injected IV. At the end of operation , the patients will be transferred to the postoperative anaesthesia care unit for routine monitoring and then to the general surgery department when they have a modified Aldrete score ≥9.

Postoperative Pain Management:

Throughout the first 24 hrs, patients will receive IV paracetamol 1 g every 8 hrs for postoperative analgesia according to the general surgery department protocol.

They also will receive IV tramadol through a patient controlled analgesia (PCA) system (concentration of 4 mg/mL); with; a 20 mg dose, a 10 mins lockout interval and a 50 mg 1 hr limit as supplementary analgesia with no background analgesia.

ELIGIBILITY:
Inclusion criteria:

* Female patients ASA II -III.
* aged 20-65 years, who will be scheduled to undergo elective unilateral breast cancer surgery.
* modified radical mastectomy.

Exclusion criteria:

* Patient refusal.
* Chronic opioid use.
* cognitive disorders.
* patients using drugs affecting the levels of calcium, phosphorus, and vitamin D, such as vitamin D supplement, calcitonin, and estrogen or its analogs, one month before enrolment.
* hyperparathyroidism or undergoing parathyroidectomy.
* diseases affecting vitamin D absorption, such as long-term diarrhea, chronic pancreatitis, biliary obstruction, colitis, partial resection of the small intestine.
* severe liver and kidney diseases.
* severe peripheral or central neuropathy.
* heart failure.
* pneumonia.
* parenteral nutrition patients.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: newly diagnosed and pathologically proven breast cancer patients who are prepared for elective breast cancer surgery will be recruited from the general surgery department of Fayoum university hospital.
Sampling Method: Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-04-20 (Actual)

PRIMARY OUTCOMES:
Incidence of moderate to severe postoperative pain | at 12 hours after surgery
  Incidence

SECONDARY OUTCOMES:
American Society of Anaesthesiologists | 24 hours before operation
  The ASA Classification is a physical status classification used to determine a patient's risk with anaesthesia1. The classification runs from ASA I to ASA VI, with the higher the number indicating a greater risk
Pain assessment by NRS | 24 hours before operation during the preoperative visit
  Pain assessment by numerical rating score (NRS) from 0 to 10 where 0 equals no pain and 10 equals the worst pain
Previous associated comorbidities | 24 hours before operation
  like hypertension, diabetes mellitus, coronary artery disease, chronic renal failure and liver impairment
Preoperative Serum 25(OH)D level (nmol/L) | 24 hours before operation
  Level
Duration of surgery | from start to the end of operation
  Duration
Total fentanyl consumption (in micrograms) | intraoperative till end of the operation
  Pain
Heart rate | baseline, every 30 minutes up to end of the operation
  measured in beats per minute
Non- invasive mean arterial blood pressure | baseline, every 30 minutes up to end of the operation
  measured in mmHg
Postoperative pain scores | at times: hour zero, hour 6, hour12, hour18, hour24 postoperative.
  NRS (Numerical rating scale) (from 0 to 10) ,0 equals no pain and 10 equals the worst pain
Total tramadol consumption | within 1st 24 hours postoperative
  measured in mg
Incidence of adverse effects | during 1st 24 hours postoperative
  nausea and vomiting (0 = no symptoms, 1 = only nausea, 2 = nausea and vomiting), respiratory depression (respiratory rate less than 10), sedation (0 = awake and alert,
  1 = quietly awake, 2 = asleep but easily arousable, 3 = deep sleep, responding to painful stimulus)
Hospital stay | from the date of the operation to the date of discharge from hospital
  in days (defined as the time elapsed from day 0; the operative day; to the time of discharge)
Patient satisfaction | up to 2 days postoperative
  will be assessed on a 4-point scale (1: excellent, 2: good 3: fair, 4: poor).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Hamed, A.professor, Principal Investigator — Faculty of medicine , Fayoum university
Locations (1):
- Fayoum university hospital, El Fayoum Qesm, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zeng X, Chen X, Li C, Shi H. Preoperative Vitamin D Level is Associated with Acute Pain After Video-Assisted Thoracoscopic Surgery: A Retrospective Cohort Study. J Pain Res. 2022 Oct 12;15:3189-3196. doi: 10.2147/JPR.S382407. eCollection 2022. PMID 36258760
- [Background] Roth DE, Abrams SA, Aloia J, Bergeron G, Bourassa MW, Brown KH, Calvo MS, Cashman KD, Combs G, De-Regil LM, Jefferds ME, Jones KS, Kapner H, Martineau AR, Neufeld LM, Schleicher RL, Thacher TD, Whiting SJ. Global prevalence and disease burden of vitamin D deficiency: a roadmap for action in low- and middle-income countries. Ann N Y Acad Sci. 2018 Oct;1430(1):44-79. doi: 10.1111/nyas.13968. Epub 2018 Sep 18. PMID 30225965
- [Background] Holick MF. Vitamin D deficiency. N Engl J Med. 2007 Jul 19;357(3):266-81. doi: 10.1056/NEJMra070553. No abstract available. PMID 17634462
- [Background] Imtiaz S, Siddiqui N, Raza SA, Loya A, Muhammad A. Vitamin D deficiency in newly diagnosed breast cancer patients. Indian J Endocrinol Metab. 2012 May;16(3):409-13. doi: 10.4103/2230-8210.95684. PMID 22629509
- [Background] Bose S, Khanna A, You J, Arora L, Qavi S, Turan A. Low serum vitamin D levels are not associated with increased postoperative pain and opioid requirements: a historical cohort study. Can J Anaesth. 2015 Jul;62(7):770-6. doi: 10.1007/s12630-015-0357-4. Epub 2015 Mar 10. PMID 25752462
- [Background] Ulitsky A, Ananthakrishnan AN, Naik A, Skaros S, Zadvornova Y, Binion DG, Issa M. Vitamin D deficiency in patients with inflammatory bowel disease: association with disease activity and quality of life. JPEN J Parenter Enteral Nutr. 2011 May;35(3):308-16. doi: 10.1177/0148607110381267. PMID 21527593
- [Background] Martinez-Alonso M, Dusso A, Ariza G, Nabal M. Vitamin D deficiency and its association with fatigue and quality of life in advanced cancer patients under palliative care: A cross-sectional study. Palliat Med. 2016 Jan;30(1):89-96. doi: 10.1177/0269216315601954. Epub 2015 Aug 27. PMID 26315460
- [Background] Sharma GN, Dave R, Sanadya J, Sharma P, Sharma KK. Various types and management of breast cancer: an overview. J Adv Pharm Technol Res. 2010 Apr;1(2):109-26. PMID 22247839
- [Background] Welsh J. Vitamin D and breast cancer: Past and present. J Steroid Biochem Mol Biol. 2018 Mar;177:15-20. doi: 10.1016/j.jsbmb.2017.07.025. Epub 2017 Jul 23. PMID 28746837
- [Background] Feldman D, Krishnan AV, Swami S, Giovannucci E, Feldman BJ. The role of vitamin D in reducing cancer risk and progression. Nat Rev Cancer. 2014 May;14(5):342-57. doi: 10.1038/nrc3691. Epub 2014 Apr 4. PMID 24705652
- [Background] Deeb KK, Trump DL, Johnson CS. Vitamin D signalling pathways in cancer: potential for anticancer therapeutics. Nat Rev Cancer. 2007 Sep;7(9):684-700. doi: 10.1038/nrc2196. PMID 17721433
- [Background] Altieri B, Grant WB, Della Casa S, Orio F, Pontecorvi A, Colao A, Sarno G, Muscogiuri G. Vitamin D and pancreas: The role of sunshine vitamin in the pathogenesis of diabetes mellitus and pancreatic cancer. Crit Rev Food Sci Nutr. 2017 Nov 2;57(16):3472-3488. doi: 10.1080/10408398.2015.1136922. PMID 27030935
- [Background] Meeker S, Seamons A, Maggio-Price L, Paik J. Protective links between vitamin D, inflammatory bowel disease and colon cancer. World J Gastroenterol. 2016 Jan 21;22(3):933-48. doi: 10.3748/wjg.v22.i3.933. PMID 26811638
- [Background] Jacobs ET, Kohler LN, Kunihiro AG, Jurutka PW. Vitamin D and Colorectal, Breast, and Prostate Cancers: A Review of the Epidemiological Evidence. J Cancer. 2016 Jan 5;7(3):232-40. doi: 10.7150/jca.13403. eCollection 2016. PMID 26918035
- [Background] Xia J, Li D, Yu G, Xu B, Gao X, Wang H, Ma Y, Li X, Xiong Y. Effects of Hypovitaminosis D on Preoperative Pain Threshold and Perioperative Opioid Use in Colorectal Cancer Surgery: A Cohort Study. Pain Physician. 2022 Oct;25(7):E1009-E1019. PMID 36288586